CLINICAL TRIAL: NCT04931420
Title: Phase II Prospective, Open-Label Randomized Controlled Trial Comparing Standard of Care Therapy With and Without Sequential Cytoreductive Interventions for Patients With Metastatic Foregut Adenocarcinoma and Undetectable Circulating Tumor-Deoxyribose Nucleic Acid (ctDNA) Levels
Brief Title: Study Comparing Standard of Care Chemotherapy With/ Without Sequential Cytoreductive Surgery for Patients With Metastatic Foregut Cancer and Undetectable Circulating Tumor-Deoxyribose Nucleic Acid Levels
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left site
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-2185
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Cancer; Foregut Carcinoid Tumor; Gastric Adenocarcinoma; Gallbladder Adenocarcinoma; Liver Cancer; GI Cancer; GI Carcinoma; Lung Cancer
Keywords: metastatic cancer; foregut cancer; metastatic foregut cancer; gastrointestinal cancer; GI cancer; cytoreductive surgery; cytoreductive treatment
MeSH Terms: conditions — Neoplasm Metastasis; Liver Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted; Thoracoscopy; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Participants Who Receive Sequential Procedures (Experimental): If you are assigned to this arm, study doctors will sequentially remove and treat all visible cancer spots with surgery, radiation, ablation, or other procedures. These interventions might include surgical removal of the diseased part of your lung, liver, lymph nodes, and/or the lining of your belly. In addition, if surgery could not be done, we could treat these diseased spots with other modalities such as radiation and/or radiofrequency/microwave ablation.
  If you're selected to be in this arm, the type of procedure you receive will vary based on your cancer and what the study doctor recommends for treatment.
  Interventions: Procedure: Video-Assisted Thoracic Surgery (VATS); Procedure: Lobectomy; Radiation: Consolidative Radiation; Radiation: Ablation Treatment; Procedure: Resection or Excision; Procedure: Peritonectomy; Other: Transarterial Radioembolization
- Arm B (Control) - Participants Who Receive Standard of Care Chemotherapy (Other): Participants in this arm receive the current standard of care chemotherapy for their specific type of gastrointestinal cancer. This treatment may include the continuation of chemotherapy and a few procedures which may improve your quality of life.
  Interventions: Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: Standard of Care Chemotherapy — * If you have cancer of the stomach or food pipe (esophagus): the preferred chemotherapy regimen includes two or three medications. These drugs include Cisplatin or Oxaliplatin and 5-fluorouracil (5 FU) in combination with Docetaxel.
  * If you have cancer of the pancreas or ampulla: the preferred chemotherapy medicines include Gemcitabine or a three-drug combination chemotherapy called FOLFIRINOX, which includes 5FU, Leucovorin, Irinotecan, and Oxaliplatin.
  * If you have bile duct cancers: a combination of Gemcitabine, platinum agents, or fluoropyrimidine will be considered.
  Arms: Arm B (Control) - Participants Who Receive Standard of Care Chemotherapy
Procedure: Video-Assisted Thoracic Surgery (VATS) — If you have lung cancer, you may receive video-assisted thoracic surgery (VATS): a type of minimally invasive thoracic surgery of the chest, performed with a thoracoscope (small videoscope) using small incisions and special instruments to minimize trauma.
  Other Names: thoracoscopy, thoracoscopic surgery or pleuroscopy,
  Arms: Arm A - Participants Who Receive Sequential Procedures
Procedure: Lobectomy — If you have lung cancer, you may receive a lobectomy:
  A major/invasive surgical procedure where an entire lobe of your lung is removed.
  Arms: Arm A - Participants Who Receive Sequential Procedures
Radiation: Consolidative Radiation — A type of radiation treatment used to kill any cancer cells that may be left in the body. It may also include a stem cell transplant or treatment with drugs that kill cancer cells.
  Other Names: intensification therapy, postremission therapy.
  Arms: Arm A - Participants Who Receive Sequential Procedures
Radiation: Ablation Treatment — Depending on the location of you cancer and the state of your cancer after chemotherapy, you may receive on the the following ablation treatments:
  -Microwave or Radiofrequency Ablation: Radiofrequency ablation (RFA) and microwave ablation (MWA) are treatments that remove liver tumors by placing a needle through the skin into the tumor. In RFA, high-frequency electrical currents are passed through an electrode in the needle, creating a small region of heat. In MWA, microwaves are created from the needle to create a small region of heat. The heat destroys the liver cancer cells.
  -General Tumor Ablation Treatment: a minimally invasive surgical method to treat solid cancers. Special probes are used to "burn" or "freeze" cancers without the usual surgery. Doctors use images of your tumor to guide where they place the needle. This requires only a tiny hole, usually less than 3 mm via which the probe is introduced.
  Arms: Arm A - Participants Who Receive Sequential Procedures
Procedure: Resection or Excision — Depending on the type of GI cancer you have and the state of your cancer after chemotherapy, you may receive a resection or excision: a surgical procedure that focuses on removing all or part of a tumor/organ/body using a sharp knife (scalpel) or other cutting instrument.
  Arms: Arm A - Participants Who Receive Sequential Procedures
Procedure: Peritonectomy — Peritonectomy is a surgery used to remove peritoneal tumors (tumors in the lining of the abdomen/stomach) from a patient. Following surgery, a heated chemotherapy bath (HIPEC) is commonly administered.
  Arms: Arm A - Participants Who Receive Sequential Procedures
Other: Transarterial Radioembolization — If you have cancer in your biliary tract (gallbladder, pancreas or liver), you may receive transarterial radioembolization known as TARE.
  TARE allows doctors to deliver radiation treatment directly to the liver using a minimally invasive technique that is designed to cause few side effects. TARE allows doctors to thread a catheter through a small incision in the participant's upper thigh through the artery that goes directly to the liver.
  Other Names: TARE
  Arms: Arm A - Participants Who Receive Sequential Procedures

SUMMARY:
This study is designed for participants who have cancer of the upper gastrointestinal (GI) tract such as cancer of the esophagus, stomach, duodenum (the initial portion of your small intestine), pancreas, bile duct (Cholangiocarcinoma), ampulla, or gall bladder with limited sites of spread (metastases). Doctors leading this study are looking to see if treating the disease using sequential procedures (more than one procedure given one after another) such as surgeries or radiation can lead to better survival and if these surgeries, combined with standard of care treatment, are safe for the treatment of upper GI cancers.

DETAILED DESCRIPTION:
This study is designed for participants who have cancer of the upper gastrointestinal (GI) tract such as cancer of the esophagus, stomach, duodenum (the initial portion of your small intestine), pancreas, bile duct (Cholangiocarcinoma), ampulla, or gall bladder with limited sites of spread (metastases).

Doctors leading this study are looking to see if treating the disease using sequential procedures (more than one procedure given one after another) such as surgeries or radiation can lead to better survival and if it is safe for the treatment of upper GI cancers.

The purpose of the proposed study is to identify a group of patients with metastatic cancer of the upper GI and biliary tract that may benefit from sequential procedures such as surgeries or radiation compared to the current standard of care chemotherapy treatment alone.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for inclusion in the study if the participant:

1. Has a newly diagnosed primary diagnosis of American Joint Committee of Cancer (AJCC) 8th Edition Stage IV esophageal or gastroesophageal adenocarcinoma, gastric adenocarcinoma, pancreatic/ampullary adenocarcinoma, intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma gallbladder adenocarcinoma, duodenal, and ampullary adenocarcinoma.

   1. All participants must have confirmed histologic diagnosis of the primary tumor
   2. Excludes patients with bone and brain metastasis (See exclusion criteria)
2. Has a primary tumor that must be locally resectable or can be treated definitively (see preferred intervention sequence). Primary tumors included are esophageal, gastric, duodenal, ampullary, pancreatic, cholangiocarcinoma, and gall bladder carcinoma. Primary tumors should be resectable or treatable with consolidative radiotherapy or ablative therapy such as microwave ablation or trans-arterial chemo/radioembolization (cholangiocarcinomas).
3. Has limited (2 sites) metastatic disease determined to be completely resectable or treatable with curative intention (see treatment algorithm) at the time of diagnosis (before induction chemotherapy). This includes:

   1. Up to 5 pulmonary metastasis amenable to wedge resection (maximum of 3 wedge resections) or lobectomy (single lobectomy) or consolidative radiation/ablative therapy
   2. Up to 5 hepatic metastasis amenable to hepatectomy (segmentectomy, sectionectomy, sectorectomy, minor hepatectomy (not more than 3 segments), wedge resection requiring a minimum of 40% of liver parenchyma following resection based on future liver remnant or a combination of partial hepatectomy and microwave ablation or trans-arterial radioembolization (TARE).
   3. Lymphatic metastases that are resectable or intervenable (limited to only two non-regional sites).
   4. Resectable peritoneal disease with a PCI of <6 and the ability to obtain a CC0 cytoreduction.
   5. Distant metastasis must be limited to two of the above-mentioned sites (a-d).
   6. If both pulmonary and liver metastasis are present (a, b), then a total of 5 lesions will be considered oligometastatic.
4. Patients with resected primary tumors can be included if they present with oligometastases at least six months after the completion of treatment of primary tumor with curative intent.
5. Has adequate organ function, as described below (Appendix 4); all screening laboratory tests should be performed within 30 days prior to the first study intervention.

   Prior Therapy
6. Patients taking substrates, inhibitors, or inducers of Cytochrome P450 3A4 (CYP3A4) should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions.

   Demographics
7. Is male or female, who is at least 18 years of age at the time of signing informed consent and less than 81 years of age at the time of signing informed consent.
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status score 0-1 at the time of randomization.

   Male Participants
9. A male participant must agree to use contraception (barrier birth control, abstinence) during the treatment period and for at least 95 days following completion, corresponding to time needed to eliminate any study intervention(s), and refrain from donating sperm during this period.

   Female Participants
10. A female participant of childbearing age is eligible to participate if she is not pregnant, not breastfeeding, and agrees to use contraception (hormonal, barrier birth control, or abstinence) for at least 95 days following completion, corresponding to time needed to eliminate any study intervention(s). Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.

    Informed Consent
11. The participant (or legally acceptable representative if applicable) provides written informed consent for the study. The participant may also provide consent for Future Biomedical Research (FBR). However, the participant may participate in the main study without participating in FBR.

Exclusion Criteria:

The participant must be excluded from the study if the participant:

Medical Conditions

1. Has a positive urine pregnancy test within 3 days prior to randomization or treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: In the event that 3 days have elapsed between the screening pregnancy test and the first dose of study intervention, another pregnancy test (urine or serum) must be performed and must be negative for the participant to start receiving study medication.
2. Has hypoxia as defined by pulse oximeter reading <92% at rest or requires intermittent or chronic supplemental oxygen.
3. Has a known additional malignancy that is progressing or has required active treatment within the past three years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
4. Has known central nervous system (CNS) metastasis and/or carcinomatous meningitis.
5. Has known osseous metastasis.
6. Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from treatment initiation, or New York Heart Association Class III or IV congestive heart failure. Medially controlled arrhythmia stable on medication is permitted.
7. Has poorly controlled hypertension defined as SBP ≥150mmHg and/or DBP ≥90mmHg.
8. Has moderate to severe hepatic impairment (Child-Pugh B or C).
9. Has a known psychiatric condition such as schizophrenia, mania, delirium, or a substance abuse disorder that would interfere with the study-related procedures.
10. Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (severe dysphasia, bowel obstruction, malabsorption).
11. Has known malignant pleural effusion or previous malignant effusion previously treated at the time of enrollment.
12. Has histologic subtypes not included in the inclusion criteria (including esophageal squamous cell carcinoma, gastroenteropancreatic neuroendocrine tumors, hepatocellular carcinoma, etc.).
13. Has ECOG performance status score 2 or greater.
14. Has a primary tumor that is not amenable to treatment.
15. Has weight loss ≥ 20% from diagnosis despite appropriate nutritional support.
16. Has progressive disease following the first three months of chemotherapy.
17. Patients with detectable circulating tumor DNA (ctDNA) following three months of induction chemotherapy.

    Prior/Concomitant Therapy
18. Has previously treated metastatic disease with surgery, radiation, or ablative procedures.

    a. Patients can be enrolled if they have received systemic chemotherapy consistent with the trial protocol, and they meet all of the inclusion criteria and none of the remaining exclusion criteria.
19. Has had major surgery within 3 weeks prior to the first dose of the study intervention. Participants must have recovered from all surgery-related complications.
20. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccine for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccine (eg. FluMist®) are live attenuated vaccines and are not allowed.

    Diagnostic Assessments
21. Has an active infection requiring systemic therapy
22. Has known active TB/ COVID infection
23. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study intervention
24. Has a known history of HIV infection
25. Has a known history of HBV (defined as HBsAg reactive) or known active HCV (defined as HCV RNA [qualitative] is detected) infection.

    Note: Testing for HBV and HCV is only required if mandated by the local health authority.

    Other Exclusions
26. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 95 days after the last study intervention.
27. Inability to receive chemotherapy and/or surgery and/or radiotherapy and/or ablative procedures due to medical/insurance reasons.
28. Has peritoneal metastases with a peritoneal carcinoma index (PCI) score of >6.
29. Requires emergency surgery due to bleeding, perforation, or obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months
  The progression free survival (PFS) of participants undergoing sequential procedures (Arm A of study) vs standard of care chemotherapy (participants in Arm B - control group) as assessed by clinical records. Progression free survival will be defined as the time from randomization to first documented disease progression or death as assessed by clinical records.

SECONDARY OUTCOMES:
6 Month Progression Free Survival | 6 months
  The percentage of participants in each arm without disease progression/death at 6 months as assessed by clinical records.
Progression Free Survival 2 | 12 months
  The percentage of participants in each arm without disease progression/death from randomization to progression on second line therapy, which includes repeat interventions.
12 Month Progression Free Survival | 12 months
  The percentage of participants in each arm without disease progression/death at 12 months as assessed by clinical records.
Median Overall Survival | 12 months
  The median overall survival of participants undergoing sequential procedures (Arm A) vs standard of care therapy (Arm B) as assessed by clinical records. Median overall survival will be defined as the time from randomization to death from any cause.
Health-Related Quality of Life | 12 months
  Health-related quality of life (HRQoL) for participants undergoing sequential procedures (Arm A) vs. the HRQoL for participants receiving standard of care treatment (Arm B). This will be assessed by quality of questionnaires completed by participants at baseline and after treatment.
Financial Toxicity | 12 months
  The financial burden and its consequences faced by participants undergoing sequential procedures vs. the financial burden experienced by participants receiving standard of care treatment (Arm B). This financial burden/toxicity will be assessed by the Comprehensive Score for Financial Toxicity (COST) questionnaire, a standardized participant-friendly questionnaire used to measure financial toxicity/burden of treatment.
Post-Procedure Morbidity of Participants in Arm A | 12 months
  The morbidity (the state of having a particular illness) of participants after undergoing sequential cytoreductive procedures (procedures used to remove tumors) as assessed by clinical records.
Post-Procedure Mortality of Participants in Arm A | 12 months
  The mortality (the number of deaths) of participants after undergoing sequential cytoreductive procedures (procedures used to remove tumors) as assessed by clinical records.
Incidence of Adverse Events Reported Among Participants in Arm B (Standard of Care Group) | 12 months
  The safety/ tolerability of standard of care treatment as assessed by reported adverse events from participants in Arm B. Adverse Events will be measured using the Common Terminology Criteria for Adverse Events (CTCAE) v.5.
Circulating Tumor DNA (ctDNA) Progression Free survival | 2 years after randomization
  The median circulating tumor DNA (ctDNA) progression free survival, which will be defined as the time from randomization to first documented disease progression, positive ctDNA detection, or death as assessed by the radiology team in participants with undetectable ctDNA. ctDNA levels in participants will be tested/assessed using liquid biopsies.
The Effect of Interventions on Circulating Tumor DNA (ctDNA) | 2 years after randomization
  The effect of interventions on circulating tumor DNA (ctDNA) levels in participants who receive aggressive interventions (Arm A) versus standard of care treatments (Arm B). The effect of interventions on ctDNA will be assessed based on recorded ctDNA levels measured using liquid biopsies at baseline and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Turaga, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: Yes